CLINICAL TRIAL: NCT04929639
Title: The Effect of Intrabdominal Pressure on Postoperative Mortality and Morbidity in Patients Undergoing Bariatric Surgery
Brief Title: The Effect of Intrabdominal Pressure in Patients Undergoing Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Other Study IDs: 09.2020.133
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Intraabdominal Pressure; Bariatrik Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: measurment of intraabdominal surgery — Immediately after intubation, while the patient is lying in the supine position, an intra-abdominal measurement will be made from the bladder catheter and recorded. Then, after the surgical site antisepsis, when the trocar required for the operation is placed by the general surgeon, another measurement will be made from the trocar port. Measurements will be recorded.

SUMMARY:
Morbid obesity is a global health problem that concerns the whole world. It is associated with many concomitant health problems such as diabetes, hypertension, congestive heart failure. There are publications showing that morbid obesity increases chronic intra-abdominal pressure, and it has been investigated that this chronic pressure exposure may cause many comorbidities accompanying obesity. When we reviewed the literature, we could not find an adequate study showing the effects of obesity-related increased intra-abdominal pressure on postoperative mortality and morbidity.

The aim of this study is to show the effect of obesity-related intra-abdominal pressure on postoperative mortality and morbidity.

DETAILED DESCRIPTION:
Our study included 80 female patients with ASA (American Society of Anesthesia) II-III, who were planned to undergo laparoscopic sleeve gasterctomy or bypass operation after ethics committee approval. BMI (body Mass Index)> 35, 18-65 years old, female, non-smoker, not undergoing revisional bariatric surgery, and not undergoing major abdominal surgery before were included. Propofol 2mg/kg, Remifentanil 1mcg/kg, and rocuronium 0.6mg/kg were administered to the patients by monitoring with ECG, pulse oximetry and non-invasive blood pressure measurement, which we performed in bariatric surgery patients in our clinic. The corrected weights of the patients were used in dose calculations as recommended by the Society of Bariatric Anesthesia. Immediately after intubation, while the patient was lying in the supine position, intra-abdominal measurement was taken from the bladder catheter and recorded. Then, after the surgical site antisepsis, when the trocar required for the operation was placed by the general surgeon, another measurement was made from the trocar port. The measurements were recorded. Arterial blood pressure, heart rate, oxygen saturation, maintenance fluids, and complications were recorded every 5 minutes intraoperatively. Postoperative hospital stay of the patients, urine output, onset time of bowel movements, and all complications were recorded.

SPSS 21.0 computer program was used for statistical analysis. The normality of the distribution of the data was evaluated with the Kolmogorov-Smirnov test. Intergroup data will be evaluated by one-way ANOVA, and in-group data will be evaluated with repetitive ANOVA test. Chi-square was used in the analysis of ordinal data. P < 0.05 will be considered as a statistically significant difference. The sample size was calculated as 80 patients at 90% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesia) II-III female patient who is planned to undergo laparoscopic sleeve gasterctomy or bypass operation will be included. BMI (body Mass Index)> 35, 18-60 years old, female, non-smoker, not undergoing revisional bariatric surgery, and not undergoing major abdominal surgery before were included

Exclusion Criteria:

* Patients with severe cardiac and respiratory distress, liver and kidney failure, and those who did not consent to the study will not be accepted into the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patient
Study Population: ASA (American Society of Anesthesia) II-III female patient who is planned to undergo laparoscopic sleeve gasterctomy or bypass operation will be included. BMI (body Mass Index)> 35, 18-60 years old, female, non-smoker
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
the effect of obesity-related intra-abdominal pressure | during procedure
  measure intra-abdominal pressure from the trochar site

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided